CLINICAL TRIAL: NCT07214220
Title: Intravascular Neuro OCT Imaging System for Aneurysm Treatment Evaluation
Acronym: INSYTE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spryte Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIP-001
Record Dates: First submitted 2025-10-01; First posted 2025-10-09 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Intracranial Aneurysm
Keywords: Intracranial aneurysm treatment; OCT
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Single arm: Use of nOCT during treatment and follow-up (Experimental): Use of nOCT during intracranial aneurysm treatment and subsequent follow-up
  Interventions: Procedure: Endovascular Intracranial aneurysm treatment; Device: nOCT imaging

INTERVENTIONS:
Procedure: Endovascular Intracranial aneurysm treatment — Endovascular Intracranial aneurysm treatment using devices such as coils, flow diverters, etc. The treatment will include devices that are all FDA approved.
Device: nOCT imaging — During the aneurysm treatment and during the subsequent follow-up, nOCT imaging will be performed.

SUMMARY:
This is an investigational study for a new medical device called the nOCT (neuro optical coherence tomography) Imaging System, which is manufactured by Spryte Medical, LLC. The nOCT Imaging System takes pictures from inside a blood vessel in your brain. These pictures give your doctor information about the inside of your blood vessel including the disease and any implanted devices.

The nOCT Imaging System consists of a probe and a console. The probe is a small, flexible wire-like device designed to navigate through catheters which have already been inserted in your body as part of your planned procedure. Catheters are small, flexible, tubes inserted in your blood vessels which allow your doctor to deliver treatments such as medications, coils, or stents directly to the affected area. The console is a unit that includes a computer, screen and laser light source. The probe is connected to the console. The console provides the probe with low-power light from the laser which is used to scan and create pictures of your blood vessel. The pictures are displayed on the screen of the console for review by your doctor and may be stored for future viewing.

The objective of the study is to evaluate the safety and effectiveness of the nOCT Imaging System to provide quality images for diagnostic assessment during endovascular intracranial aneurysm treatment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

Subject age ≥ 18 and ≤ 75 years

Subject has a pre-procedure mRS ≤ 3

Subject is undergoing a planned treatment for an intracranial aneurysm, unruptured or ruptured

Subject understands the investigational procedure, consents to participation, is willing to comply with study follow-up requirements and provides a signed informed consent document

Parent artery has a diameter ≥ 1.3 mm and ≤ 6.0 mm as measured by angiography.

Exclusion Criteria:

Subjects with a minimum platelet count of < 100,000/μL.

Subjects who have suffered an ischemic stroke or transient ischemic attack within the past 30 days.

Subject has an acutely ruptured aneurysm with a Hunt & Hess score ≥ 4

Subject has an infectious, blister-like, fusiform, dissecting, traumatic or mycotic aneurysm confirmed by angiography

Subject has challenging anatomy that in the investigator's opinion is not suitable for safe delivery of an 0.021" catheter, including stenosis > 70% or excessive tortuosity

Subject presents with other medical or surgical co-morbidities limiting his/her life expectancy to less than one year

Subject is, in the opinion of the investigator, unlikely to comply with the study protocol or follow-up requirements.

Subject with any condition which in the opinion of the treating physician would place the subject at an elevated risk of embolic stroke

Subject with known allergy or other contraindication to heparin, iodinated contrast, or dual-antiplatelet medication

Subject has ipsilateral carotid or vertebral artery stenosis greater than 50%

Subject underwent stenting, angioplasty, or endarterectomy procedures of an extracranial (carotid or vertebral artery) or intracranial artery within 30 days prior to treatment.

Subject has serious concurrent medical conditions including bacteremia or sepsis, acute renal failure at the time of the procedure, and major coagulation system abnormalities that in the opinion of the investigator could significantly increase risk

Subject has severe intracranial vasospasm not responsive to medical therapy

Subject has chronic kidney disease stage ≥ 4 and is not undergoing dialysis

The subject is pregnant or breastfeeding at the time of admission or plans to become pregnant during their participation in the trial

Subject is currently participating in another clinical research trial involving an investigational device or drug

Subject is under judicial protection or legal guardianship

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-07-07 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Safety - Adverse Events | peri-procedural
  All peri-procedural adverse events (AE) from the index procedure.
Effectiveness | peri-procedural
  Image quality, defined as clear image length (CIL) for images obtained during the index procedure.

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing plans are under evaluation pending sponsor policy and regulatory guidance